CLINICAL TRIAL: NCT07344532
Title: The Effect of Preoperative Abdominal Superficial Effleurage Training on the Development of Postoperative Constipation in Patients Undergoing Abdominal Surgery
Brief Title: Effect of Preoperative Abdominal Effleurage on Postoperative Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mehmet Ozkeskin, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOzkeskin7126
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Constipation; Abdominal Surgery; Postoperative Constipation
Keywords: Postoperative Constipation; Abdominal Surgery; Abdominal Effleurage; Non-Pharmacological Intervention
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group receiving preoperative abdominal superficial effleurage training in addition to routine care or a control group receiving routine care only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abdominal Superficial Effleurage Group (Experimental): Participants in this group will receive preoperative training on abdominal superficial effleurage in addition to routine clinical care. Following surgery, patients will perform the effleurage technique for approximately five minutes, one to three times daily, during periods without pain.
  Interventions: Behavioral: Abdominal Superficial Effleurage Training
- Control Group (No Intervention): Participants in the control group will receive routine clinical care only and will not receive abdominal superficial effleurage training during the study period.

INTERVENTIONS:
Behavioral: Abdominal Superficial Effleurage Training — Abdominal superficial effleurage is a gentle abdominal massage technique involving stroking movements from the right upper quadrant toward the left lower quadrant of the abdomen. Participants will be trained preoperatively to perform the technique, which will take approximately five minutes per session and will be performed one to three times daily postoperatively during pain-free periods.
  Arms: Abdominal Superficial Effleurage Group

SUMMARY:
This randomized controlled study aims to evaluate the effect of preoperative abdominal superficial effleurage training on the development of postoperative constipation in patients undergoing abdominal surgery. Participants will be randomly assigned to an intervention group receiving abdominal superficial effleurage training in addition to routine care or to a control group receiving routine care only. The effleurage technique will be taught preoperatively and performed by patients postoperatively. Postoperative constipation will be assessed on the 10th postoperative day using the Bristol Stool Form Scale. The findings of this study are expected to contribute to non-pharmacological nursing interventions for the prevention of postoperative constipation.

DETAILED DESCRIPTION:
Postoperative constipation is a common complication following abdominal surgery and may negatively affect patient comfort, recovery, and quality of life. Non-pharmacological nursing interventions that support bowel motility are therefore of increasing interest in perioperative care. Abdominal superficial effleurage is a gentle massage technique applied to the abdominal surface and is thought to stimulate intestinal peristalsis and promote bowel function.

This prospective, randomized controlled study will be conducted with patients scheduled to undergo abdominal surgery. A total of 42 patients will be randomly assigned to either the intervention group (n=21) or the control group (n=21) using a computer-generated randomization method. Patients in the intervention group will receive preoperative training on abdominal superficial effleurage in addition to routine clinical care, while patients in the control group will receive routine clinical care only. To minimize interaction between groups, data from the control group will be collected prior to the intervention group.

Abdominal superficial effleurage will be taught during the preoperative period and performed by patients postoperatively. The technique involves gentle stroking movements starting from the right upper quadrant of the abdomen and progressing toward the left lower quadrant. Each session will last approximately five minutes and will be performed one to three times daily during periods when the patient is not experiencing pain. Postoperative constipation will be evaluated on the 10th postoperative day through a telephone interview using the Bristol Stool Form Scale. Study data will be analyzed using appropriate descriptive and inferential statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo abdominal surgery
* Patients who are able to communicate verbally
* Patients who agree to participate in the study and provide written informed consent

Exclusion Criteria:

* Patients with preoperative constipation
* Patients with known gastrointestinal diseases affecting bowel motility
* Patients who are unable to perform abdominal superficial effleurage
* Patients with cognitive impairment or communication difficulties
* Patients who refuse to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-09-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Constipation | 10 days postoperatively
  Postoperative constipation will be assessed using the Bristol Stool Form Scale through a telephone interview conducted on the 10th postoperative day. Stool types 1 and 2 will be considered indicative of constipation.

SECONDARY OUTCOMES:
Stool Consistency | 10 days postoperatively
  Stool consistency will be evaluated using the Bristol Stool Form Scale (BSFS), a 7-point validated scale ranging from Type 1 (separate hard lumps, indicating severe constipation) to Type 7 (watery, no solid pieces, indicating severe diarrhea). Higher scores indicate looser stool consistency and a tendency toward diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Ozkeskin, PhD, Principal Investigator — Ege University

IPD SHARING:
Plan to Share IPD: No